CLINICAL TRIAL: NCT03035253
Title: A Phase 1b Study of OMP-305B83 Plus FOLFIRI or FOLFOX as Second Line Therapy in Subjects With Metastatic Colorectal Cancer
Brief Title: A Study of OMP-305B83 in Subjects With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B83-003
Record Dates: First submitted 2016-12-22; First posted 2017-01-27 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — navicixizumab; Antibodies, Bispecific; IFL protocol; Folfox protocol

ARMS (1):
- OMP-305B83 combined with FOLFIRI or FOLFOX (Experimental)
  Interventions: Drug: OMP-305B83; Drug: FOLFIRI; Drug: FOLFOX

INTERVENTIONS:
Drug: OMP-305B83
  Other Names: bispecific monoclonal antibody
Drug: FOLFIRI — Treatment will consist of OMP-305B83 and the FOLFIRI chemotherapy regimen.
Drug: FOLFOX — Treatment will consist of OMP-305B83 and the FOLFOX chemotherapy regimen.

SUMMARY:
The purpose of this study is to test the safety and efficacy of an experimental drug, OMP-305B83, when given in combination with FOLFIRI or FOLFOX. OMP-305B83 is a humanized bispecific monoclonal antibody and was developed to target cancer stem cells. Based on preclinical studies, it is believed that OMP-305B83 may block the growth of cancer stem cells and may also impair the productive growth of new blood vessels, which tumors need to grow and spread.

The study is sponsored by OncoMed Pharmaceuticals, which is referred to as OncoMed or the Sponsor.

DETAILED DESCRIPTION:
This is an open-label, Phase 1b dose escalation and expansion study of OMP-305B83 plus FOLFIRI or FOLFOX to evaluate the safety, efficacy, and pharmacokinetics of OMP-305B83 in combination with FOLFIRI or FOLFOX in patients with metastatic Colorectal Cancer. This study consists of a screening period, a treatment period, and a post-treatment follow-up period in which patients will be followed for survival for up to 5 years. Patients will be enrolled in two stages: a dose-escalation stage and an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1
* Age >21 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ and marrow function
* For women of childbearing potential and men with partners of childbearing potential, agreement (by patient and/or partner) to use two effective forms of contraception from study entry through at least 6 months after the termination visit.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Receiving any other investigational agents or any other anti-cancer therapy
* Receiving prior hepatic intra-arterial chemotherapy
* Known significant clinically significant gastrointestinal disease
* Patients with brain metastases (treated or untreated) leptomeningeal disease, uncontrolled seizure disorder, or active neurologic disease
* Significant intercurrent illness that will limit the patient's ability to participate in the study or may result in their death over the next 18 months
* Pregnant or nursing women
* Inability to comply with study and follow up procedure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | Subjects will be treated and observed for DLT through the end of the first cycle (Days 0-28).
  The maximum tolerated dose (MTD) or maximum administered dose (MAD) will be determined in patients treated with OMP-305B83 in combination with FOLFIRI or FOLFOX

SECONDARY OUTCOMES:
Safety of OMP-305B83 in combination with FOLFIRI or FOLFOX will be assessed by adverse event monitoring, physical exams, vital signs, clinical laboratory testing, ECGs, echocardiograms, anti-OMP-305B83 testing, and subject interview on an ongoing basis. | Through study completion, an average of 8 months
Immunogenicity (in terms of formation of anti-drug antibod(ies) against OMP-305B83 in percentage of subjects) of OMP-305B83 in combination with FOLFIRI or FOLFOX | Through study completion, an average of 8 months
Response Rate assessed by RECIST criteria 1.1 | At 56 day intervals while on treatment, through study completion, an average of 8 months
Response Rate assessed by tumor marker CEA | At 28 day intervals while on treatment, through study completion, an average of 8 months
Progression Free Survival | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Cancer Care & Hematology - Fort Collins, Fort Collins, Colorado
  - University of Michigan Health System, Ann Arbor, Michigan
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah